CLINICAL TRIAL: NCT06252272
Title: Generation of Organotypic Liver Cultures for the Identification of Biomarkers for the Prevention and Treatment of Liver Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RS1822/23
Record Dates: First submitted 2024-01-17; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Non-pharmacological study of a biological nature, low level interventional prospective intervention for the preparation of cultures of organotypic liver slices (hLSC)
Masking Description: Biopsy sample in an area of liver macroscopically free from parenchymal alterations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy sample in an area of liver macroscopically free from parenchymal alterations (Other): Patients undergoing abdominal surgery for primary or secondary liver tumors (liver metastases from colorectal, pancreatic, or breast), from which we proceed to the preparation of organotypic cultures of liver (hLSC) derived from liver biopsies taken from patients undergoing abdominal surgery for primary or secondary liver tumors for the molecular characterization of liver fibrosis.
  Interventions: Diagnostic Test: Biopsy from patients undergoing surgery abdominal.

INTERVENTIONS:
Diagnostic Test: Biopsy from patients undergoing surgery abdominal. — A small portion (about 10 mm in diameter) of liver tissue was collected macroscopically free from alterations of the parenchyma obtained in the open at the site surgery for primary or secondary liver tumors, for the preparation of cultures of organotypic liver slices.

SUMMARY:
Low-level, interventional, biological and non-pharmacological study prospective intervention for the preparation of organotypic human liver slice cultures Liver Slice Culture (hLSC) applying the protocol described by Jiang and collaborators.

DETAILED DESCRIPTION:
Human liver slice culture hLSCs will be used from non-tumor liver tissue collected by biopsy from patients undergoing abdominal surgery, who have signed informed consent and agree to perform a liver biopsy for the specific research protocol.

The study is "low level interventional" when a small portion (approximately 10 mm in diameter) of liver tissue macroscopically free from parenchymal alterations obtained in the open at the site of surgery for primary or secondary liver tumors will be taken (hepatic metastases from colorectal, pancreatic or breast cancer). The goal is to create organotypic liver cultures (hLSC) derived from liver biopsies taken from patients undergoing abdominal surgery.

for primary or secondary liver tumors for the molecular characterization of liver fibrosis.

Use hLSC to study the liver microenvironment and molecular determinants involved in fibrosis through single cell sequencing; compare the sequencing data obtained with hLSC with that obtained via characterization of a GEMM whose generation is foreseen in the same project financed by the MoS.

To generate this GEMM, the pro-fibrotic Hipk2 gene was specifically deleted in the tissue liver (HIPK2-liver knock-out, HIPK2-LKO) and liver fibrosis will be induced through a high-fat, low-choline diet.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old;
* patients for whom it is indicated to undergo abdominal surgery for tumors primary or secondary liver diseases;
* patients who express informed consent to the study.

Exclusion Criteria:

* medical contraindication to performing a liver biopsy;
* liver cirrhosis;
* macroscopic signs of chronic liver disease;
* moderate or severe steatosis;
* cholestasis;
* hepatic necrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Molecular characterization of liver fibrosis | 24 months
  Creation of organotypic cultures of liverderived from liver biopsies taken from patients undergoing abdominal surgery for primary or secondary liver tumors for the molecular characterization of liver fibrosis.Patients will undergo abdominal surgery (as per clinical practice), during which a biopsy will be performed in an area of the liver macroscopically free from parenchymal alterations, approximately 20/25 slices will be obtained from each sample. The hLSCs will come used to study the hepatic microenvironment in the presence or absence of pro-fibrinogenetic stimuli e of anti-fibrotics by time-lapse analysis and confocal immunofluorescence microscopy multiple and through single cell sequencing.

SECONDARY OUTCOMES:
Study of the hepatic microenvironment | 24 months
  Use hLSCs to study the liver microenvironment and the molecular determinants involved in it fibrosis through single cell sequencing (single-cell RNA sequencing);
Compare the sequencing data | 24 months
  Compare the sequencing data obtained with hLSCs with those obtained through the characterization of a GEMM. A biopsy will be performed after abdominal surgery (as per clinical practice), in an area of the liver macroscopically free from parenchymal alterations.
  hLSCs will be analyzed over the following week for viability and fibrosis induction using fibrosis-specific stains for time-lapse dynamic imaging (IncuCyte), i.e. picrosirius red, Masson's trichrome, and quantitative RT-PCR and multiplex immunofluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Soddu, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy